CLINICAL TRIAL: NCT06692478
Title: Benefits of Intrahospital Exercise Program in Pediatric Hematopoietic Stem Cell Transplant-A Randomized Control Trial
Brief Title: Benefits of Intrahospital Exercise Program in Pediatric HSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16-127
Record Dates: First submitted 2017-11-02; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-04

CONDITIONS: Hematopoietic Stem Cell Transplant; Pediatric Cancer; Deconditioning
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The physical therapist doing the evaluations, the data analyst, and primary investigator will all be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): This structured exercise program will incorporate a specially designed, low intensity, resistance based exercise regime created by our physical therapist. In addition to standard of care, it consists of strengthening, endurance, stretching and relaxation exercises tailored according to age and their ability to perform activities throughout their hospitalization. This exercise program will be done three times a week for 30-45 mins supervised by the same physiotherapist throughout hospitalization and will be self-administered every weekend. A home exercise program printout with the appropriate resistance exercises will be provided to the family upon discharge, with instructions on how often to complete throughout the week. Discharged children will attend one supervised exercise session per week with the physiotherapist for six weeks. The family and patient will also be provided a weekly sheet to check off the days they completed strengthening and endurance exercises.
  Interventions: Behavioral: Exercise regimen
- Standard of Care (No Intervention): The second arm of the study involves patients following standard of care during the HSCT period in the hospital with PT evaluation and management prescribed as needed by their transplant medical team including any additional PT interventions as a result of clinical indications. No additional intervention is incorporated in this group

INTERVENTIONS:
Behavioral: Exercise regimen — Age 4-6 years: Target lower extremity, core and upper extremity strengthening and activity tolerance. With supervision by the PT, the patient will walk in their room, and complete the following through play: squat, single leg stance, climb onto couch, half kneel to stand, quadruped and tall kneeling.
  Age 7-21 years: First component will be strengthening exercises completed in bed or on a mat while sitting or standing. Multiple levels of exercises will be available, so that the program can be tailored to each patient and to their ability to perform activities. The exercises included will focus on core, hip musculature, and upper extremity strengthening; including exercises in quadruped and prone positioning, as well as supine, sitting and standing. Thera-Band will be used to increase resistance as needed. The second component will be endurance. Since the patients will be confined to their room this will include ambulation within the room, recumbent or pedal exerciser and step ups.
  Arms: Exercise

SUMMARY:
This randomized control study examines the effect of an intrahospital exercise regimen on the physical deconditioning that occurs due to hematopoietic stem cell transplant in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 4-21 years of age who present for hematopoietic stem cell transplant.
2. Karnofsky (if ≥16 years) or Lansky (if <16 years) score >60 at enrollment and prior to each testing point
3. Parental/guardian permission (informed consent) and child assent prior to transplant.

Exclusion Criteria:

1. Patients with any preexisting need for gait assistance such as crutches, wheelchair, braces, or walker
2. Previous stem cell transplant in the last 6 months
3. Patients with grade 3 or greater sensory/motor neuropathy

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline 6-minute walk test at 6 weeks discharge. | Average of 100 days post-transplant
  Test of Endurance (Pre-transplant, at discharge, and 6 weeks discharge.)
Change from Baseline Manual Muscle Testing at 6 weeks post discharge | Average of 100 days post-transplant
  Muscle strength
WeeFIM | Average of 100 days post-transplant
  Change from Baseline Functionality at 6 weeks post discharge.

SECONDARY OUTCOMES:
PROMISE Measures | Average of 100 days post transplant
  Change from Quality of Life measurements based off of physical, mental, and social categories at 6 weeks post discharge
Time Out of Bed | through study completion, average of 1 year
  Log of average time out of bed for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
IPD on request